CLINICAL TRIAL: NCT04939207
Title: Improving the Cost-effectiveness of Coronary Artery Disease Diagnosis
Brief Title: Safety and Cost-efficiëncy of New Imaging Techniques in Patients Suspected of Coronary Artery Disease
Acronym: iCORONARY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); UMC Utrecht (Other)
Responsible Party: Principal Investigator, Martin J. Swaans, Principal investigator, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL7739.100.21; 852002131 (Other Grant/Funding Number: ZonMW)
Record Dates: First submitted 2021-06-07; First posted 2021-06-25 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Angina pectoris; Coronary arteriosclerosis; CT scan; Cardiac catheterization; Coronary angiography; Myocardial fractional flow reserve
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris | interventions — Angiography

STUDY DESIGN:
Intervention Model Description: After coronary CT-scan, patients will be randomized in one of three possible study arms. One arm will receive additional CT-derived calculation of coronary blood flow, one arm will receive angiography-derived calculation of coronary blood flow and one arm will receive standard routine care. Standard care consists of coronary angiography and invasive coronary blood flow measurements. The results of these tests determine the need for treatment of coronary artery disease. After these tests, patients will be treated and followed according to routine care guidelines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- CT-derived FFR (Experimental): In this study arm, the need for coronary revascularization will be determined by CT-derived Fractional Flow Reserve (FFR) calculations
  Interventions: Diagnostic Test: CT-FFR
- Angiography-derived FFR (Experimental): In this study arm, the need for coronary revascularization will be determined by FFR-calculations derived from angiographic images
  Interventions: Diagnostic Test: Angiography-derived FFR
- Routine Care (Active Comparator): In this study arm, the need for coronary revascularization will be determined by angiography and invasive FFR-measurements
  Interventions: Diagnostic Test: Angiography with invasive FFR-measurements

INTERVENTIONS:
Diagnostic Test: CT-FFR — CT-images will be processed by an algorithm to calculate FFR-values of the full coronary tree
  Arms: CT-derived FFR
Diagnostic Test: Angiography-derived FFR — FFR-values are calculated during coronary angiography based on the acquired images of the coronary arteries
  Arms: Angiography-derived FFR
Diagnostic Test: Angiography with invasive FFR-measurements — during coronary angiography, a specialized pressure wire is passed through the coronary stenosis to calculate FFR based on the difference between the actual pressure and the expected pressure in the hypothetical healthy coronary artery.
  Arms: Routine Care

SUMMARY:
Yearly, 180 000 patients in the Netherlands are referred to a cardiologist with symptoms suspected of coronary artery disease (CAD). To assess this, multiple diagnostic tests are available. Non-invasive imaging tests, such as coronary CT-scan, are safe, relatively cheap and can effectively rule-out CAD. However, when CAD is present, coronary CT-scan cannot assess the restriction in blood flow caused by the stenosis. Cardiac angiography with invasive blood flow measurements is required to assess this restriction in blood flow. This is an invasive test, more expensive than CT and it is accompanied by certain risks.

Most patients in whom CAD is present do not need treatment, and would therefore benefit from non-invasive diagnostic tests. To reduce the number of unnecessary cardiac angiography with flow measurements, new imaging techniques have been developed. These techniques use CT- or angiographic images to calculate the restriction in coronary blood flow and determine the need for treatment. This study is designed to assess the safety and efficacy of these techniques when used as an addition to coronary CT-scan.

Subjects are eligible if their CT-scan indicates possibly significant CAD. To determine need for treatment of a subject's CAD, the investigators will randomize subjects in three arms. One arm consists of additional CT-derived calculation of coronary blood flow, one arm consists of angiography-derived calculation of coronary blood flow and one arm consists of standard care, coronary angiography and invasive coronary blood flow measurements. After these tests, subjects are treated and followed according to routine care guidelines. Additionally, subjects are requested to complete 5 questionnaires in a 12 month follow-up period.

The investigators expect that the total number of invasive cardiac angiographies with additional blood flow measurements can be reduced by half with the use of new imaging techniques. The investigators expect that this will lead to a reduction in healthcare costs, complications and a lower burden of diagnostic tests for patients. The investigators do not expect a difference in primary endpoints between the study groups.

DETAILED DESCRIPTION:
Only a small proportion of the 180 000 patients that are referred to a cardiologist each year in the Netherlands with complaints of angina pectoris or shortness of breath suffer from coronary stenosis in such a degree that revascularisation is required. To identify these patients, multiple diagnostic tests are available. Simple non-interventional imaging tests, such as coronary CT-scan, are safe, relatively cheap and can effectively rule-out coronary artery disease. However, when coronary artery disease is present, coronary CT-scan cannot assess the restriction in blood flow caused by the stenosis. Cardiac angiography with invasive blood flow measurements is required to assess this restriction in blood flow. This is an invasive test, more expensive than CT and it is accompanied by certain risks.

In retrospect, many patients unnecessarily undergo cardiac angiography with, if deemed neccessary, flow measurements. These patients do not need treatment for coronary artery disease. To reduce the number of unnecessary cardiac angiography with flow measurements, new imaging techniques have been developed. These techniques use CT- or angiographic images to calculate the restriction in coronary blood flow and determine the need for treatment. These new imaging techniques have been tested extensively in observational studies. Currently, there is no consensus in the optimal diagnostic pathway resulting in major differences in strategies between hospitals. Moreover,data on cost-effectiveness is lacking.

This study is designed to assess the safety and efficacy of these techniques when used as an addition to coronary CT-scan. Our target population will be patients with complaints of angina pectoris or shortness of breath for which the patients will undergo coronary CT-scan. If the CT-scan shows one or more possibly flow-limiting stenoses, further diagnostic testing is required. These subjects are randomized in one of three possible arms. One arm will receive additional CT-derived calculation of coronary blood flow, one arm will receive angiography-derived calculation of coronary blood flow and one arm will receive standard care. Standard care consists of coronary angiography and invasive coronary blood flow measurements. The results of these tests determine the need for treatment of coronary artery disease. After these tests, subjects are treated according to routine care guidelines. Subjects are requested to complete 5 questionnaires in a 12 month follow-up period. The primary endpoint is a composite of MACE - all-cause mortality, aborted sudden cardiac death, myocardial infarction and unplanned hospitalization for chest pain leading to urgent revascularization during the 12-month follow-up period. Secondary endpoints consist of cost-effectiveness, the number of avoided invasive coronary angiographies and flow measurements and quality of life. The investigators will use hospital patient files and completed questionnaires to collect information about events during the follow-up period until the last included subject has completed their final questionnaire.

The investigators expect that the total number of invasive cardiac angiographies with additional blood flow measurements can be reduced by half with the use of new imaging techniques. The investigators expect that this will lead to a reduction in healthcare costs, complications and a lower burden of diagnostic tests for patients. The investigators do not expect a difference in primary endpoints between the study groups.

In addition to the randomised controlled trial, all eligible subjects whose coronary CT-scan does not show possibly significant coronary artery disease (CAD-RADS 0-2) are included in a patient registry. Because of absent or limited coronary artery disease, additional diagnostic testing is not needed in these patients. These subjects are requested to answer 5 questionnaires in a 12-month period, similar to the subjects included in the RCT-part of the trial. The outcome measures of this part of the trial are similar to those of the RCT. Our primary outcome is the occurrence of MACE-events, secondary outcomes are quality of life and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* The subject is willing and able to provide informed consent and adhere to study rules and regulations and follow-up
* The subject is clinically suspected of having (recurrent) angina pectoris or an equivalent and suspected coronary artery disease, based on symptoms and signs, history, clinical examination and baseline diagnostic testing (e.g. ECG recording and laboratory tests) as described in the 2019 ESC guideline on chronic coronary syndromes.
* The subject has had ≥64 multidetector row coronary CTA or will undergo coronary CTA as part of usual care deemed by the treating physician with ≥64 multidetector row coronary CTA.

Exclusion Criteria:

* The subject is suffering from unstable angina pectoris.
* The subject is suffering from decompensated congestive cardiac failure.
* The subject is suffering from a known non-ischemic cardiomyopathy.
* The subject has a history of PCI or CABG.
* The subject has had pacemaker or internal defibrillator leads implanted.
* The subject has a prosthetic heart valve.
* There is a severe language barrier.
* The subject participates in any other clinical trial that interferes with the current study.
* Clinical condition prohibiting subsequent interventional therapy as indicated by the results of the imaging procedures.
* The subject is or might be pregnant.
* The subject does not comply or is not able to comply to the imaging guidelines for the performance and acquisition of CCTA by the Society of Cardiac Computed Tomography (SCCT), including:

  * The subject is suffering from a cardiac rhythm other than sinus rhythm.
  * The subject is morbidly obese (Body Mass Index (BMI) > 40).
  * The subject is not able to sustain a breath-hold for 25 seconds.
  * The subject is unable to remain in supine position for at least 30 minutes.
  * The subject has known allergies to or contra-indications to receiving an iodinated contrast agent. Contraindications to receiving an iodinated contrast agent: Glomerular Filtration Rate (GFR) < 45 ml/min/1,73m2 and if the subject is diabetic or has at least two risk factors for developing contrast induced renal failure a GFR < 60 ml/min/1,73m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 825 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Safety of non-invasive imaging techniques | 12 months
  The number of Major adverse cardiovasculare events (MACE) as all-cause mortality, aborted sudden cardiac death, myocardial infarction and unplanned hospitalization for chest pain leading to urgent revascularization in a 12 month follow-up period.

SECONDARY OUTCOMES:
Cost-effectiveness | 12 months
  Calculated using the total costs of the initial diagnostic tests, any additional tests or treatments for coronary artery disease, hospital admissions for suspected cardiac events and other costs that can be attributed to possible coronary artery disease. The medical costs will be calculated by the use of imta Medical Cost Questionnaire (iMCQ). Cost-effectiveness will be calculated by combining the total costs with the productivity loss using the iMTA Productivity Cost Questionnaire (iPCQ)
Seattle Angina Pectoris Questionnaire | 12 months
  This questionnaire focuses on the presence of and limits caused by angina pectoris symptoms
PHQ-9 Questionnaire | 12 months
  The Patient Health Questionnaire focuses on the mental health of the subject
PROMIS-10 Questionnaire | 12 months
  This questionnaire focuses on the overall health care consumption of the subject
Avoided coronary angiographies | 12 months
  To determine the fraction of avoided Cardiac Angiography's measurement by the use of CT-FFR. This is done by substracting the number of subjects in the CT-FFR group that received invasive angiography during the follow-up period from the total number of subjects in the CT-FFR group. Without the use of CT-FFR, all subjects in this group would have received invasive coronary angiography.
Avoided invasive FFR-measurements | 12 months
  To determine the fraction of avoided FFR measurement by the use of angiography-derived FFR-calculations. This is done by substracting the number of subjects in het angiography-based FFR-group that received invasive FFR-measurements during the follow-up from the total number of subjects in the angiography-based FFR-group that would have received invasive FFR-measurements based on their angiographic views if angiography-based FFR would not have been available. Many of the subjects in this group would have received invasive FFR-measurements if angiography-based FFR would not have been available.

CONTACTS AND LOCATIONS:
Overall Officials: Martin J Swaans, Dr., Principal Investigator — St. Antonius Ziekenhuis Nieuwegein; Tim Leiner, Prof. Dr., Principal Investigator — UMC Utrecht
Locations (4):
- Netherlands (4):
  - Catharina Hospital, Eindhoven, North Brabant
  - Maasstad Hospital, Rotterdam, South Holland
  - St. Antonius Hospital, Nieuwegein, Utrecht
  - UMC Utrecht, Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, the data will be locally saved at the st. Antonius Hospital and can be made available at request for reuse in other studies.
Supporting Information: Study Protocol, SAP
Time Frame: After publishing the main study articles, raw and modified data can be made available at request
Access Criteria: These criteria will be made in consultation with the legal advisor of our institution and have not yet been drafted.
  Specific degrees in the field of research have to be demonstrated, as wel as links with hospitals or research institutes of the researcher/physician (e.g. an employee contract)

REFERENCES:
- [Derived] Peper J, Becker LM, Bruning TA, Budde RPJ, van Dockum WG, Frederix GWJ, Habets J, Henriques JPS, Houthuizen P, Mohamed Hoesein FAA, Planken RN, Voskuil M, Bots ML, Leiner T, Swaans MJ. Rationale and design of the iCORONARY trial: improving the cost-effectiveness of coronary artery disease diagnosis. Neth Heart J. 2023 Apr;31(4):150-156. doi: 10.1007/s12471-023-01758-3. Epub 2023 Jan 31. PMID 36720801